CLINICAL TRIAL: NCT05924087
Title: Interventional Therapy of Tracheal Stenosis After Percutaneous Tracheotomia
Brief Title: Interventional Therapy of Tracheal Stenosis
Status: Recruiting | Type: Observational
Sponsor: Asklepios Neurological Clinic Bad Salzhausen (Other)
Responsible Party: Sponsor
Other Study IDs: ITTS10_06_2023
Record Dates: First submitted 2023-06-10; First posted 2023-06-29 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Tracheal Stenosis Following Tracheostomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
After respiratory weaning, decannulation is sought. To do this, the tracheal cannula is first unblocked, so that patients no longer breathe in and out through the cannula, but (at least partially) "passing" the cannula by the natural route. In the presence of tracheal stenosis there is increased breathing effort, possibly restlessness and stridor. This constellation of symptoms suggests the suspicion of tracheal stenosis, so in the next step a tracheoscopy is performed to confirm or exclude tracheal stenosis. In case of symptomatic tracheal stenosis and at least 30-50% stenosis of the trachea (clinical symptoms can be expected from a 30-50% stenosis) then appropriate therapy (here: cryotherapy, other techniques only in exceptional cases) is planned. The goal is to be able to remove the tracheal cannula (long term) after successful therapy, so that patients do not have to be permanently provided with a tracheal cannula. There is no definitive/evidence-based standard therapy for the treatment of tracheal stenosis. Cryotherapy is a gentle therapy that has already been applied and described for the treatment of tracheal stenosis (see above). The examination is performed as part of an analgesic dose, as is routine for a bronchoscopy (in-house SOP). After treatment, a follow-up is planned for about 10 days later.

ELIGIBILITY:
Inclusion Criteria:

* Tracheal stenosis after percutaneous tracheotomy.

Exclusion Criteria:

* Pregnant or breast-feeding women of childbearing potential who refuse pregnancy test.
* lack of consent to participate in the study.
* surgical tracheotomy.
* Involvement of the larynx (above the first tracheal brace).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients after successfull respiratory weaning with symptomatic trachealstenosis
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Decannulation | 12 months
  Rate of successful decannulations after intervention up to discharge from inpatient treatment.

SECONDARY OUTCOMES:
Technical success | 12 months
  technical success of the intervention (endoscopically not clinically relevant tracheal stenosis).
Reintervention(s) | 12 months
  Number of interventions required.
Type of intervention | 12 months
  Type of intervention(s) (cyroablation, APC, loop extraction).
Clinical success | 12 months
  Clinical success (no stridor, no dyspnoea).
Additional treatment | 12 months
  Number of patients requiring surgical treatment/stent.

CONTACTS AND LOCATIONS:
Locations (1):
- Neurologische Klinik Bad Salzhausen, Nidda, Germany